CLINICAL TRIAL: NCT02133352
Title: Proof of Concept Study of Ranolazine in the Treatment of Pulmonary Hypertension Associated With Diastolic Left Ventricular Dysfunction
Brief Title: Study of Ranolazine in the Treatment of Pulmonary Hypertension Associated With Diastolic Left Ventricular Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30217
Record Dates: First submitted 2014-05-06; First posted 2014-05-08 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Hypertension; Diastolic Left Ventricular Dysfunction
Keywords: pulmonary hypertension; diastolic dyfunction
MeSH Terms: conditions — Hypertension, Pulmonary; Ventricular Dysfunction, Left | interventions — Ranolazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ranolazine (Experimental): Ranolazine- initiated at 500mg twice daily and increased to 1000mg twice daily as tolerated after 2wks; the tolerated dose will be used for the remainder of the Treatment Period.
  Interventions: Drug: Ranolazine

INTERVENTIONS:
Drug: Ranolazine — Single arm- ranolazine, initiated at 500 mg BID and increased to 1000 mg BID as tolerated
  Other Names: Ranexa

SUMMARY:
This is a single center, open-label trial designed to assess the safety and efficacy of ranolazine (Ranexa) in patients with pulmonary hypertension associated with left ventricular diastolic dysfunction. All patients will receive active drug. The study includes a screening period, 6 month treatment period and a follow up period. Eligible patients who provide informed consent and who meet all inclusion/exclusion criteria will be enrolled in this study.

There is neither proven therapy for patients with diastolic dysfunction-associated pulmonary hypertension nor for patients with diastolic dysfunction alone. Ranolazine, an inhibitor of cardiac repolarization (sodium channels), could represent a new and effective treatment of this entity.

DETAILED DESCRIPTION:
This single center, prospective, open-label trial to assess the safety and efficacy of ranolazine in subjects with pulmonary hypertension associated with left ventricular diastolic dysfunction includes a screening period, 6 month treatment period and a follow up period. Eligible subjects who provide informed consent and who meet all inclusion/exclusion criteria will be enrolled in this study. All subjects will receive active study drug. There is no placebo group or use of control subjects. Treating will begin with 500mg twice daily and increased to 1000mg twice daily as tolerated after 2wks; the tolerated dose will be used for the remainder of the Treatment Period. Ranolazine will be limited to 500 mg BID in patients taking moderate inhibitors of CYP3A, including diltiazem, verapamil, aprepitant, erythromycin, fluconazole, grapefruit juice or grapefruit-containing products. During the Treatment Period subjects will be provided bottles of study medication to take home. Throughout the Treatment Period, subjects will return to the clinic for safety and/or efficacy assessments as well as resupply of Study Medication. Once the Treatment Period is complete, subjects will return to the clinic for a Follow-Up visit 14 days after the last dose of study medication, for a final safety assessment. Other therapies or possibly extension of the ranolazine treatment may be considered after completion of the Treatment Period at the discretion of the Investigator and will be recorded at the follow-up visit. Subjects who continue taking ranolazine (as part of there clinical care), will be asked to return for a 1 year follow up visit for safety and efficacy assessments.

As part of Amendment 2 (submitted November 2013), subjects who continue on ranolazine after the 6 month treatment period (as part of their clinical care) will be asked to return for further follow-up testing to better assess the safety and efficacy of the drug. The visit can be conducted once the patient has been on drug for a total of one year or greater (including the 6 month treatment period). This would replace the 1 Year follow-up visit for subjects who have not yet completed the visit and will be an additional visit for those subjects who have.

Subjects can opt to continue on ranolazine regardless of if they agree to complete the Post Treatment Follow up visit. They do not have to continue with the study after the treatment phase has been completed in order to stay on ranolazine. The PI and study personnel will complete the required forms for the Ranexa Connect application if patient wishes to stay on drug. The Ranexa Connect Program assists patients in obtaining insurance coverage of ranolazine and financial assistance if needed.

This is a 6 month, single center, prospective, open-label trial. All subjects will be receiving active treatment, ranolazine at doses approved by the FDA. Subjects will begin treatment at 500mg twice daily and increase to 1000mg twice daily as tolerated after 2 weeks. Subjects will take study drug twice daily with or without food. Ranolazine will be limited in subjects taking CYP3A including diltiazem, verapamil, arprepitant, erythromycin, fluconazole, grapefruit juice or grapefruit juice containing products. The study will consist of 3 periods: a screening period, a treatment period, and a follow-up period.

Subjects will be asked to come to the study center for 9-10 visits over the course of 6 months. Other therapies or possibly extension of the ranolazine treatment may be considered after completion of the treatment period at the discretion of the Investigator at the follow up visit. Subjects who continue on ranolazine after completion of the treatment period of the study will be asked to return for follow up testing.

ELIGIBILITY:
Inclusion Criteria:

* Written consent prior to any study procedure
* Men or women, ages 18 to 75 years
* Suspicion of Pulmonary Hypertension by echo (RVSP ≥ 50mmHg) or diagnosis of Pulmonary Hypertension by cardiac cath (mPAP ≥25 mmHg at rest)
* LVEF ≥50%, (by ECHO, radionuclide imaging, or cardiac cath)
* 6MWT distance ≥150m and ≤450m at both time points within the Screening Period
* NYHA/WHO functional class II-III
* RHC measurements on Study Day 1: 1) mean pulmonary artery pressure (MPAP) ≥25 mmHg; 2) pulmonary artery occlusion pressure (PAOP) ≥18 mmHg and ≤30 mmHg; 3) pulmonary artery diastolic pressure (PADP) - PAOP ≤10 mmHg

Exclusion Criteria:

* Presence or history of any of the following cardiovascular co-morbidities or conditions: Hypotension at Screening (defined as a resting SBP≤90mmHg). Hypertension at Screening (defined as resting SBP ≥200mmHg), Unstable cardiovascular disease including paroxysmal atrial fibrillation or unstable angina, Amyloidosis, hypertrophic obstructive cardiomyopathy, restrictive cardiomyopathy, or constrictive pericarditis, History of myocardial infarction, coronary artery bypass graft surgery, or percutaneous cardiac intervention, Significant valvular heart disease, Cerebrovascular accident or transient ischemic attack
* Exercise tolerance limited by non-cardiac causes (exercise-induced asthma, malignancy, obesity, musculoskeletal disorder).
* Clinically significant psychiatric, addictive (DSM-IV criteria), neurologic disease or condition that would compromise his/her ability to give informed consent, participate fully in this study, or prevent adherence to the protocol
* Any other condition or co-morbidity that, in the opinion of the Investigator, would compromise his/her ability to give informed consent, participate fully in this study, or prevent adherence to the protocol
* Clinically significant laboratory abnormalities, including: Positive Hep B surface antigen or Hep C antibody, Positive HIV test within one year of Study Day 1, Serum alanine aminotransferase (ALT) ≥ 2.0 x ULN, Total bilirubin ≥ 1.2 x ULN (unless evidence of Gilbert's syndrome). Serum creatinine ≥ 2.5mg/dL (or calculated creatinine clearance less than or equal to 30mL/min). Hemoglobin less than or equal to 10g/dL (subject may qualify for the study following diagnosis and treatment of anemia, if the anemia is due to iron and/or vitamin deficiency).

Patients with moderate or severe hepatic impairment (Child-Pugh Classes B or C) or requiring hemidialysis.

* Subject has received any other investigational medication within the 30 days prior to Screening
* Prior treatment with ranolazine
* Pregnancy or lactation
* Women of childbearing potential and men without vasectomies who are not using barrier method of contraception
* Subject has the presence, or history, of malignancy that required significant medical intervention within the preceding 3 months and/or is likely to result in death within the next 2 years (exception of basal cell, non-metastatic squamous cell carcinoma of the skin, and carcinoma in-situ of the cervix)
* Treatment for pulmonary hypertension with epoprostenol (Flolan), treprostinil (Remodulin), iloprost (Ventavis), bosentan (Tracleer), ambrisentan (Letairis), sildenafil (Revatio), tadalafil (Adcirca). The use of sildenafil, tadalafil, or vardenafil is prohibited for any reason within 7 days of hemodynamic assessments on Days 1 and 180).
* Patients with QTc > 500 msec at baseline
* Treatment with potent CYP3A inhibitors, including ketoconazole, itraconazonle, clarithromycin, nefazodone, nelfinavir, indinavir, & saquinavir
* Treatment with CYP3A inducers, including rifampin, rifabutin, rifapentin, phenobarbital, phenytoin, carbamazepine, and St. John's wort.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-07; Primary Completion 2013-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harrison Farber, MD, Principal Investigator — Boston University
Locations (1):
- Boston University Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ranolazine: Ranolazine- initiated at 500mg twice daily and increased to 1000mg twice daily as tolerated after 2wks; the tolerated dose will be used for the remainder of the Treatment Period.
  Ranolazine: open label/Single arm- ranolazine, initiated at 500 mg BID and increased to 1000 mg BID as tolerated
Period: Main Study (180 Day)
Arm/Group | Ranolazine
Started | 10
Completed | 10
Not Completed | 0
Period: Longer Term Extension
Arm/Group | Ranolazine
Started | 10
Completed (4 of the initial 10 subjects agreed/consented to participate in the longer term extension) | 4
Not Completed | 6
Not completed — 4 of the initial 10 subjects agreed/cons | 6

BASELINE CHARACTERISTICS:
Arm/Group | Ranolazine
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (6.1)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in mPAP, PAOP and Pulmonary Vascular Resistance (PVR)
Description: Assess the percent change in mPAP, PAOP and pulmonary vascular resistance (PVR) by RHC.
  Additional RHC completed at optional follow up for patients remaining on ranolazine upon completion of 180 day period.
Time Frame: 180 days
Population: We hypothesize that patients with pulmonary hypertension associated with diastolic left ventricular dysfunction treated with Ranolazine (initiated at 500 mg twice daily and increased to 1000mg twice daily) would have improved hemodynamic parameters, functional capacity and exercise tolerance compared to baseline.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Ranolazine
Number analyzed (Participants) | 10
percentage change
  % Change in mPAP | -21 (7.43)
  % Change in PAOP | -39 (7.28)
  % Change in PVR | -4.0 (153.86)

2. Secondary Outcome: Percent Change in Other Hemodynamic Parameters
Description: Assess % change in other hemodynamic parameters, by RHC, from baseline afeter 180 days of ranolazine.
  Right atrial pressure (RAP) Systolic pulmonary artery pressure (SPAP) Diastolic pulmonary artery pressure (DPAP) Cardiac output (CO) Cardiac index (CI)
Time Frame: 180 days
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ranolazine
Number analyzed (Participants) | 10
percent change
  RAP | -56 (4.59)
  SPAP | -12 (11.41)
  DPAP | -33 (5.79)
  CO | 22 (1.78)
  CI | 24 (0.87)

3. Secondary Outcome: 6 Minute Walk Test (6MWT)
Description: Assess the change from baseline in 6 minute walk test (6MWT) after 180 days of twice daily ranolazine Optional follow up for some patients also includes 6MWT.
Time Frame: 180 days
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Ranolazine
Number analyzed (Participants) | 10
meters | 33.7 (35.17)

4. Secondary Outcome: Change in Cardiac Size and Function
Description: Assess changes from baseline in measurements of cardiac size and function obtained by MRI after 180 days of twice daily ranolazine.
  An additional MRI may be completed at optional follow up visit for patients continuing on ranolazine following completion of the 180 day treatment period.
Time Frame: 180 days
Measure: Mean (Standard Deviation); unit: % ejection fraction
Arm/Group | Ranolazine
Number analyzed (Participants) | 5
% ejection fraction
  RVEF | 3 (.88)
  LVEF | 5.4 (.2)

5. Secondary Outcome: Change in Echocardiogram Parameters (LVEF)
Description: To assess the changes from baseline in echocardiographic parameters (left ventricular geometry and function, LVEF, evidence of diastolic dysfunction, SPAP, right ventricular geometry and function, degree of tricuspid regurgitation) after 180 days of twice daily ranolazine.
  An additional echo may be completed at optional follow up visit for patients continuing on ranolazine following completion of the 180 day treatment period.
Time Frame: 180 days
Measure: Mean (Standard Deviation); unit: LVEF %
Arm/Group | Ranolazine
Number analyzed (Participants) | 6
LVEF % | .67 (1.9)

6. Secondary Outcome: Change in BNP Cardiac Biomarker
Description: Assess the change from baseline in BNP cardiac biomarkers after 180 days of twice daily ranolazine.
  Cardiac biomarkers may be completed at optional follow up visit for patients continuing on ranolazine following completion of the 180 day treatment period.
Time Frame: 180 days
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ranolazine
Number analyzed (Participants) | 10
pg/mL | 32.1 (5.2)

ADVERSE EVENTS:
Time Frame: 180 Days
Arm/Group | Ranolazine
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranolazine (N=10)
Bradycardia with junctional ventricular escapes (Cardiac disorders) | 1 (1) — Hospital admission revealing bradycardia with ventricular escapes.
GI bleed (Gastrointestinal disorders) | 1 (1) — Patient admitted for GI bleed. Felt to be unrelated to study drug.
CHF Exacerbation (Cardiac disorders) | 1 (1) — Patient admitted 02Jan2013, resolved 12Jan2013. Unrelated to study drug.
Chest pain (Cardiac disorders) | 1 (1) — Patient admitted with chest pain on 07APR2013. Not thought to be related to drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranolazine (N=10)
diarrhea (Gastrointestinal disorders) | 1 (1)
increased shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
difficulty concentrating (General disorders) | 1 (1)
patient fall (General disorders) | 1 (1)
worsening foot pain/gout (Immune system disorders) | 1 (1)
common cold (General disorders) | 4 (7)
increased stomach discomfort (Gastrointestinal disorders) | 1 (1)
urinary tract infection (Infections and infestations) | 1 (1)
lightheadedness (General disorders) | 3 (4)
elevated blood sugar (Endocrine disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 3 (4)
increased fatigue (General disorders) | 1 (1)
sore throat (General disorders) | 1 (1)
muscle spasm (General disorders) | 1 (1)
kidney infection (Infections and infestations) | 1 (1)
intermittent increased back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
buttocks/upper leg pain (General disorders) | 1 (1)
thumb pain (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size; not all subjects completed Day 180 assessments

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No